CLINICAL TRIAL: NCT06044454
Title: RADICAL: A Mixed Methods Study to Assess the Clinical Effectiveness and Acceptability of an Artificial Intelligence Software to Prioritise Chest X-ray (CXR) Interpretation
Brief Title: Radiograph Accelerated Detection and Identification of Cancer in the Lung
Acronym: RADICAL
Status: Active, not recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Qure.ai Technologies Pvt. Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: INGN23RM028; 23/NW/0211 (Other: Ethics Committee)
Record Dates: First submitted 2023-08-29; First posted 2023-09-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Service deployment: Intervention Chest X-ray received - care team (standard of care) CT scan - care team (standard of care)
  Interventions: Other: qXR

INTERVENTIONS:
Other: qXR — a software product that uses artificial intelligence to triage, prioritise, and (for tuberculosis only) diagnose based upon identified abnormalities within the CXR.

SUMMARY:
Lung cancer is the most common cause of cancer death in the UK yet compared to Europe it has low survival rates.The NHS aims to find 75% of cancers at an early stage as this can improve the chances of survival.

To support this target, Qure.ai have developed the UK-approved qXR product, which is a software program that automatically analyses chest x-rays using artificial intelligence to identify features associated with lung cancer, indicative of other diagnoses, or that contain no abnormal features ('normal'). qXR is a class IIb medical device that can be used by radiologists to prioritise reporting based upon the presence or absence of these features. This may improve the accuracy and efficiency of reporting these images.

The project includes different elements including:

i) Clinical effectiveness study across 3 sectors within NHS Greater Glasgow and Clyde (NHSGGC).The primary objective is to assess the clinical effectiveness of qXR to prioritise patients that have suspected lung cancer (identified from AI analysis of a chest x-ray) for follow-on CT.

Primary study outcome measure - Time to 'decision to recommend CT', or to a decision not to undertake CT for CXR acquired with USC (CXR acquired to CXR reported).

Secondary objectives include:

i) To assess the potential utility of qXR within the optimised lung cancer pathway in terms of the impact on both patient treatment and radiological workflow.

ii) A technical evaluation utilising retrospective and prospective cohorts. The technical retrospective study will determine the performance of qXR using a sample of 1000 CXR images from all chest x-ray referral sources across all sectors (this differs from the prospective study, which only examines outpatient referred chest x-rays).

iii) A health economic evaluation. Use of per patient healthcare utilisation costs to model cost benefits of qXR, including implementation of supported reporting of normal CXR.

iv) A qualitative evaluation to assess acceptability and barriers to scale-up and implementation

DETAILED DESCRIPTION:
A clinical effectiveness study will be conducted in 3 NHS Greater Glasgow and Clyde sectors over a 12-month period.

Sectors will be identified and initiated into the qXR solution with a 30 day implementation period. The order in which sites will receive the qXR intervention will be determined by computer-based randomisation.

The technical retrospective study will determine the performance of qXR using a sample of 1000 CXR images from all chest x-ray referral sources across all sectors (this differs from the prospective study, which only examines outpatient referred chest x-rays). An economic evaluation will be conducted comparing costs and outcomes with and without the introduction of qXR. The software potentially impacts costs via two mechanisms: the identification of normal can enhance efficiency of CXR reporting; and the identification of USCs can support the prioritisation of CXRs that show signs of lung cancer, accelerating the provision of CT, which leads to faster diagnosis and treatment, and ultimately better outcomes.

Qualitative evaluation: To determine acceptability, staff interviews and patient focus groups will be carried out.

Data will be collected by an experienced qualitative researcher using a semi-structured interview guide, developed based on the key constructs of the Theoretical Framework of Acceptability. All interviews will be conducted via Zoom at a mutually agreed upon date and time and are estimated to last, on average, around 45 minutes.

To capture the NHS service user perspective, the investigators will also conduct three online focus groups with approximately 20 NHS service users.

ELIGIBILITY:
Inclusion Criteria:

* Unconsented patients ≧ 18 years old with frontal chest radiograph, acquired consecutively during usual care through the outpatient (including GP) referral pathway only, whose radiograph has not already been reported (applies to clinical effectiveness and health economic evaluation studies).
* Unconsented patients ≧ 18 years old with frontal chest radiograph, sampled from images already acquired and reported in the current or previous calendar year (applies to technical evaluation).
* Key stakeholders such as NHS service users, healthcare staff and NHS management (applies to qualitative evaluation).

Exclusion Criteria:

* Patient has requested that they are removed from the study, or has objected to the use of AI in their routine clinical care and this has been subsequently upheld by the health board (applies to clinical effectiveness study, health economic evaluation and technical evaluation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Service deployment within a single health board (NHS Greater Glasgow and Clyde), within the following sectors and hospitals:
  Clyde Sector
  * The Royal Alexandra Hospital
  * Inverclyde Royal Hospital
  * Vale of Leven Hospital
  South Sector
  * Queen Elizabeth University Hospital
  * New Victoria Hospital
  * Gartnavel General Hospital
  * West Glasgow Ambulatory Care Hospital
  North Sector
  * Glasgow Royal Infirmary
  * Stobhill Hospital
  At each participating site, the investigators will identify all patients referred through the outpatient pathway (including GP-referrals). This will include those with suspected lung cancer referred for CXR.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Time to 'decision to recommend CT', or to a decision not to undertake CT for CXR acquired with USC (CXR acquired to CXR reported) | through study completion, an average of 1 year
  Time to 'decision to recommend CT', or to a decision not to undertake CT for CXR acquired with USC (CXR acquired to CXR reported)

SECONDARY OUTCOMES:
Time from acquisition to reporting of all CXRs | through study completion, an average of 1 year
  Time from acquisition to reporting of all CXRs
Time to diagnosis of lung cancer | through study completion, an average of 1 year
  Time to diagnosis of lung cancer
Time to treatment initiation lung cancer | through study completion, an average of 1 year
  Time to treatment initiation lung cancer
Number of hospital visits during screening pathway | through study completion, an average of 1 year
  Number of hospital visits during screening pathway
Hospitalisation within 6 and 12 months CXR acquisition | through study completion, an average of 1 year
  Hospitalisation within 6 and 12 months CXR acquisition
Death within 6 and 12 months of CXR acquisition | through study completion, an average of 1 year
  Death within 6 and 12 months of CXR acquisition
Percentage of CXRs not identified by qXR as suspected lung cancer that the radiologist refers for CT for USC | through study completion, an average of 1 year
  Percentage of CXRs not identified by qXR as suspected lung cancer that the radiologist refers for CT for USC
Percentage of non-USC that are referred for CT with subsequent detection of lung cancer | through study completion, an average of 1 year
  Percentage of non-USC that are referred for CT with subsequent detection of lung cancer
Model performance e.g. sensitivity, specificity, positive and negative predictive values. | through study completion, an average of 1 year
  Model performance e.g. sensitivity, specificity, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: David Lowe, Principal Investigator — NHS Greater Glasgow and Clyde Board HQ
Locations (4):
- United Kingdom (4):
  - Glasgow Royal Infirmary (North Sector), Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Queen Elizabeth University Hosp (South Sector), Glasgow
  - The Royal Alexandra Hospital (Clyde Sector), Paisley

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duncan SF, McConnachie A, Blackwood J, Stobo DB, Maclay JD, Wu O, Germeni E, Robert D, Bilgili B, Kumar S, Hall M, Lowe DJ. Radiograph accelerated detection and identification of cancer in the lung (RADICAL): a mixed methods study to assess the clinical effectiveness and acceptability of Qure.ai artificial intelligence software to prioritise chest X-ray (CXR) interpretation. BMJ Open. 2024 Sep 20;14(9):e081062. doi: 10.1136/bmjopen-2023-081062. PMID 39306349